CLINICAL TRIAL: NCT01800851
Title: Calorimetry, Insulin Resistance and Energy Metabolism Study to Understand the Risk of Obesity in Kidney Transplanted Patients
Acronym: CALIMERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Laboratoire Régional de Nutrition Humaine (Other); Hopital Gabriel Montpied (Other); Agrément pour la Recherche Biomédicale n°03047S (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CHU-0146; 2007-A00287-46
Record Dates: First submitted 2013-02-15; First posted 2013-02-28 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Renal Failure; Kidney Transplantation; Weight Gain; Insulin Resistance; Diabetes
Keywords: Kidney transplantation; Energy expenditure; Weight gain; Insulin resistance
MeSH Terms: conditions — Kidney Failure, Chronic; Weight Gain; Insulin Resistance; Diabetes Mellitus

ARMS (3):
- no weight gain (Experimental): The characteristics of the renal transplant patients are compared with those of 10 healthy volunteers matched for age and lean body mass
  Interventions: Other: Energy expenditure evaluation in calorimetric chamber
- weight gain (Experimental): The characteristics of the renal transplant patients are compared with those of 10 healthy volunteers matched for age and lean body mass
  Interventions: Other: Energy expenditure evaluation in calorimetric chamber
- lean body mass (Other): The characteristics of the renal transplant patients are compared with those of 10 healthy volunteers matched for age and lean body mass
  Interventions: Other: Energy expenditure evaluation in calorimetric chamber

INTERVENTIONS:
Other: Energy expenditure evaluation in calorimetric chamber

SUMMARY:
Weight gain is a common complication after transplantation. It has adverse effects such as hypertension, dyslipidemia, and insulin resistance. Weight gain is implicated in the increased cardiovascular risk and the long-term loss of graft function. Weight loss achieved by a suitable dietary intervention in these patients transplanted kidney can correct lipid disorders and facilitate balance blood pressure. The identification of mechanisms responsible for weight gain would suggest prevention strategies and allow to align the caloric energy needs of renal transplant patients.

DETAILED DESCRIPTION:
Weight gain is a common complication after transplantation. It has adverse effects such as hypertension, dyslipidemia, and insulin resistance. Weight gain is implicated in the increased cardiovascular risk and the long-term loss of graft function. Weight loss achieved by a suitable dietary intervention in these patients transplanted kidney can correct lipid disorders and facilitate balance blood pressure. The identification of mechanisms responsible for weight gain would suggest prevention strategies and allow to align the caloric energy needs of renal transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* Male patient, affiliated to a social security system
* Aged 35 to 65 years
* Renal transplant for more than a year and less than 6 years
* Treated by anticalcineurin
* Patient stopped all treatment with corticosteroids for more than 3 months
* Patient with stable renal function defined by a calculated creatinine clearance between 30 and 90 mL/min/1, 73m according to the Cockcroft and Gault
* Written informed consent after detailed explanation of the protocol.
* Increase in body weight of at least 3kg during the two years prior to the inclusion of 10 patients. Stable or increasing weight less than 1kg for 10 other patients.
* HIV and HCV serology negative

Exclusion Criteria:

* Female patients
* Diabetic (type 1 or type 2) before transplantation or patients who developed diabetes after transplantation and requiring anti-diabetic treatment at the time of inclusion
* Obese patient at the time of transplantation, as defined by a body mass index> 30%
* Multiple kidney transplant or other organ transplant the kidney
* Patient with lower limb edema, congestive heart failure, and/or uncontrolled hypertension.
* Patient with a change in body weight> 3 kg in the last 3 months
* Patient with an infection 3 months before inclusion
* Subjects infected with hepatitis B, hepatitis C virus or human immunodeficiency
* Patient with acute rejection within 3 months prior to inclusion
* Patient not treated by anticalcineurin
* Patient with a modification of immunosuppressive therapy within 3 months prior to inclusion
* Patient with unstable psychiatric condition
* Patient smoking> 5 cigarettes / day
* Alcoholic patient (unweaned)
* Patient with stage 4 renal failure (<30 mL/min/1, 73m ²) and stage 5 (<15 mL/min/1, 73m ²)
* hemodialysis patient
* Patient with acute renal failure defined by a 25% increase in creatinine within 3 months prior to inclusion
* Person under guardianship or not subject to social security
* Person in period Exclusion File National Healthy Volunteers
* Person who refuses to give his written consent to participation

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | at day 1

SECONDARY OUTCOMES:
Body composition | at day 1
Food intake | at day 1
Estimation of physical activity | at day 1
Insulin resistance | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Elisabeth HENG, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France